CLINICAL TRIAL: NCT06113757
Title: Investigation of Efficacy and Safety of Electrical Signal Therapy Provided by Dr Biolyse® Device in COVID-19 Disease: Prospective, Controlled Medical Device Clinical Trial
Brief Title: Investigation of Efficacy and Safety of Electrical Signal Therapy Provided by Dr Biolyse® Device in COVID-19 Disease
Acronym: DoBiC-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AVB Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASA02-005
Record Dates: First submitted 2023-10-31; First posted 2023-11-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: COVID-19 Pneumonia; Virus Diseases; COVID-19
Keywords: electrification; signal therapy; dr.biolyse
MeSH Terms: conditions — Virus Diseases; COVID-19

STUDY DESIGN:
Intervention Model Description: The clinical study is designed on a comparative control basis, comparing treatment interventions applied to patients. As there are no medical devices with antiviral effects, the comparison is structured to evaluate the progression and effects of the disease. It is specifically designed to compare the change between the group receiving only liquid serum support and supportive treatment and the group receiving Dr. Biolyse® treatment, with the aim of demonstrating the development and impact of the disease.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dr.Biolyse (Experimental): When you join the Dr. Biolyse® Therapy Group, you will be given electrical signal therapy with the Dr. Biolyse® device. Before the application, the area where the electrodes will be cleaned with appropriate solutions. In addition, 500-1000 ml of isotonic serum will be supplemented according to your weight, just before the first electrical signal application during the day. The treatment protocol to be applied to DBTG patients consists of device therapy and daily fluid support therapy. No medication or different device applications are performed.
  Interventions: Device: Signal Therapy provided by Dr.Biolyse device; Other: Liquid Support Treatment
- Kontrol (Experimental): In the CG patients, who constitute the Comparison Group, the same non-drug fluid support therapy applied in device therapy will be repeated (isotonic, isolated 500 ml). As both groups of patients will receive fluid support therapy, the impact of the device on the disease will be observed with monitored parameters.
  Interventions: Other: Liquid Support Treatment

INTERVENTIONS:
Device: Signal Therapy provided by Dr.Biolyse device — Before the application, the area where the electrodes will be cleaned with appropriate solutions. In addition, 500-1000 ml of isotonic serum will be supplemented according to your weight, just before the first electrical signal application during the day. Electrical signal will be applied to the lung and upper leg area for 90 minutes in the morning, noon, and evening on the first 3 days, 60 minutes in the morning and evening on the 4th and 5th days, to the lung and upper leg area. During your first hospitalization, blood will be drawn from you daily for 5 days and evaluated in terms of various biochemical parameters and detailed molecular analyzes.
  Other Names: Quantum Signal Therapy Technology
  Arms: Dr.Biolyse
Other: Liquid Support Treatment — The control group will only receive fluid therapy and will be monitored with the same blood parameters throughout the hospitalization.

SUMMARY:
Dr. Biolyse® is a device with artificial intelligence that works in sync with the immune system and can be integrated like an element of this system. It is designed to develop chemical immunity within the body against infections. It gives electrical signals to the body without causing any pain and suffering to the patient. The electric current it applies is of a type that is not used in homes, and it is the frequency feature of direct current.

The aim of this study is to evaluate the safety and efficacy of the Biolyse device. for minimizing the use of drugs in COVID-19 patients and treating drug-related organ damage during treatment We hope that by conducting this study, we will obtain sufficient data to obtain approval (CE certification) for routine use and marketing of this medical device in patients. Once this happens, we will be able to ensure that this device is accessible/usable for patients suffering from similar diseases, especially COVID-19, regardless of any studies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-65
* Patients with mild moderate complicated or uncomplicated COVID 19 pneumonias
* Those who accept to be followed up and treated as an inpatient
* Those who have at least one laboratory and clinical finding that can be evaluated during follow-up

Exclusion Criteria:

* Patients with severe course or COVID 19 pneumonia requiring intensive care follow-up
* Pregnant or breastfeeding women
* Epilepsy, Arrhythmia, Dementia, heart failure, severe lung disease, patients with active malignancy and those with pacemaker
* "Vulnerable Population" patients defined in ICU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Reaction | 5 days, during hospital stay
  The fundamental principle of this study is to prioritize the preservation of the volunteer's health. Therefore, in the event of multiple serious adverse effects that pose a threat to the life of the volunteers during device applications and cannot be prevented, or if the device applications fail to achieve the targeted effectiveness within the framework of the examined parameters, the research will be terminated.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Chairman of the Board, Principal Investigator — AVB Biotech A.S.
Locations (1):
- Bezmialem Vakif University Dragos Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ustunova S, Haciosmanoglu E, Bulut H, Elibol B, Kilic A, Hekimoglu R, Tunc S, Atmaca R, Kaygusuz I, Tunc S, Tunc GB, Meral I. A low direct electrical signal attenuates oxidative stress and inflammation in septic rats. PLoS One. 2021 Sep 9;16(9):e0257177. doi: 10.1371/journal.pone.0257177. eCollection 2021. PMID 34499695
- See also: A low direct electrical signal attenuates oxidative stress and inflammation in septic rats — https://pubmed.ncbi.nlm.nih.gov/34499695/